CLINICAL TRIAL: NCT02126904
Title: Comparison of the Time to Recurrence After Ranibizumab or Aflibercept Loading for Age-related Macular Degeneration
Brief Title: Comparison of the Time to Recurrence Between Ranibizumab and Aflibercept
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yokohama City University Medical Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Maiko Inoue, Associate Professor, Yokohama City University Medical Center
Other Study IDs: 1310006
Record Dates: First submitted 2014-04-27; First posted 2014-04-30 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-04

CONDITIONS: The Injection Burden

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- IVR group
  Interventions: Drug: IVA group

INTERVENTIONS:
Drug: IVA group

SUMMARY:
The investigators compared the time to recurrence after ranibizumab or aflibercept loading in patients with AMD.

ELIGIBILITY:
Inclusion Criteria:

* They must have had BCVA better than 20/400 and had three consecutive induction treatment of ranibizumab or aflibercept.

Exclusion Criteria:

* patients with eye diseases that could potentially influence the visual acuity of the studied eye, such as glaucoma, macular hole, diabetic retinopathy, or rhegmatogenous retinal detachment.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients were treated at Yokohama City University Medical Center between January 2012 and October 2013.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Time to recurrence after induction phase | More than 3 months from baseline
  Time frame depends on patients because recurrence time is different.

CONTACTS AND LOCATIONS:
Locations (1):
- Yokohama City University Medical Center, Yokohama, Kanagawa, Japan